CLINICAL TRIAL: NCT05856318
Title: Preconception to pOst-partum Study of Cardiometabolic Health in Primigravid PregnancY
Brief Title: Cardiometabolic Health in First Time Pregnancy
Acronym: POPPY
Status: Recruiting | Type: Observational
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Collaborators: University of Cambridge (Other); University of Bristol (Other); University College, London (Other); King's College London (Other); Imperial College London (Other); St George's, University of London (Other); University of Glasgow (Other); Wellcome Trust (Other)
Responsible Party: Principal Investigator, Dr Ian B Wilkinson, Head of Division, Division of Experimental Medicine & Immunotherapeutics, Cambridge University Hospitals NHS Foundation Trust
Other Study IDs: POPPY
Record Dates: First submitted 2023-04-17; First posted 2023-05-12 (Actual); Last update posted 2024-04-09 (Actual); Status verified 2024-04

CONDITIONS: Cardiometabolic Health; Pregnancy Related; Diabetes; Placental; Syndrome, Dysfunction; Heart Diseases
Keywords: cardiometabolic; pregnancy; diabetes; childbirth; placental syndrome; heart disease; nulliparous; CVD risk; cardiovascular
MeSH Terms: conditions — Diabetes Mellitus; Syndrome; Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Urine, Umbilical Cord
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pregnancy ~3000 participants: Actively planning to conceive within approximately 12 months of study registration. No previous pregnancies.
- Non-Pregnancy ~500 participants: Not planning to conceive within 18 months of study registration. No previous pregnancies.

SUMMARY:
Women who experience placental complications (syndromes) during pregnancy, such as pre-eclampsia (high blood pressure and kidney problems), gestational hypertension (high blood pressure during pregnancy) and fetal growth restriction (baby being small) have twice the risk of developing heart disease and diabetes later in life, compared to women who have a healthy pregnancy.

This study aims to assess risk factors for heart disease and diabetes in women who are actively trying to conceive, before and during their pregnancy, and 9-12 months after delivery of their baby, to see whether placental syndromes make a difference to their heart health. This will allow us to understand, if, and how, placental syndromes increase the risk of heart disease and diabetes, and, therefore, how best to reduce this risk and potentially prevent placental syndromes in the future. The investigators will also recruit women who are NOT planning pregnancy, as a control group.

DETAILED DESCRIPTION:
Pre-eclampsia (PE), gestational hypertension (GH) and fetal growth restriction (FGR) share a common aetiology in that they arise from complex interactions between defective placentation, trophoblast dysfunction and the maternal cardiovascular and other systems. These placental syndromes affect approximately one in five nulliparous women and are a leading cause of maternal and child morbidity. Although usually considered self-limiting, and cured by delivery, placental syndromes are associated with an increased risk of maternal hypertension, diabetes and cardiovascular disease (CVD) in later life. Indeed, as summarised by NICE, PE is associated with a 4-fold increased risk of hypertension, and 2-fold excess risk of ischaemic heart disease and stroke. Similarly, Danish National Registry data show that women with GH have a 6-fold risk of subsequent hypertension, a 3-fold risk of diabetes and a 2-fold risk of CVD; similar to that reported for PE.

Whilst these risks have most impact in later life, they are evident almost immediately - women who develop hypertension in pregnancy have a 12 to 25-fold risk of developing permanent hypertension in the year after giving birth, compared to women with a normotensive pregnancy. Approximately one third of women in their 40s who had a hypertensive pregnancy, develop hypertension over the subsequent decade, compared with only 11% who had a normotensive pregnancy. Precursors of CVD (i.e. pre-clinical phenotypes) are also apparent in the early post-partum period in women who experience a placental syndrome. Increased aortic stiffness, elevated carotid intima-media thickness (cIMT) and left ventricular dysfunction have all been reported in women with previous PE/GH and FGR.

Whether placental syndromes simply "unmask" women with pre-existing (pre-conception) poor cardiometabolic health, or cause later maternal diabetes and CVD, remains unknown. If the former is correct, then improving cardiometabolic health in young women prior to conception could be key to reducing the incidence of placental syndromes. Conversely, if placental syndromes lead to CVD and diabetes independently of established cardiometabolic risk factors (e.g. by causing end organ damage), a focus on CVD/diabetes prevention in this high-risk group of women is likely to reduce the burden of these diseases. To date, studies with pre-conception measures of cardiometabolic risk factors are few, modest in patient number and detail, and have yielded conflicting results.

The study will test definitively, the hypothesis that placental syndromes adversely affect cardiometabolic health post-partum, independently of women's pre-conception cardiometabolic health. To do this, an observational, prospective study of healthy, nulliparous women, recruited pre-pregnancy will be undertaken.

Recruitment of the study population will utilise local advertisements and networks, social media and charitable organisations involved in pregnancy research. The study focus is nulliparous women to maximize the occurrence of placental syndromes (risk is highest in first pregnancies), and to remove any confounding effect of previous pregnancies.

The study does not involve randomisation of participants; participant study arm will be determined by individuals and their intention to conceive during the determined study period, or not, in line with the inclusion/exclusion criteria.

A sufficient number of women will be recruited to the Pregnancy arm of the study to yield 1500 viable pregnancies (~3000 women, based on our feasibility data). Of these, the investigators anticipate that 135 women will experience a placental syndrome, taking into account attrition. A Non-Pregnancy study arm, women voluntarily planning not to conceive during their involvement in the study; n~500 will also be recruited, to act as a control arm.

Individual participant study duration will last between approximately 12 and 33 months dependent on study arm and timings around pregnancy and follow-up. For those in the Non-Pregnancy arm study duration will last approximately 18 months, ending after the second follow up visit. Study duration for those in the Pregnancy arm will vary, between 12 months and 33 months, dependent on time from recruitment to pregnancy occurrence and/or occurrence of placental syndrome; those (Pregnancy arm) participants who do not become pregnant will experience a shorter study duration (12 months) and only a proportion of those experiencing a healthy pregnancy will attend a final follow-up visit 18 months after delivery.

The output of this study will primarily aim to determine to what extent the association between placental syndromes and maternal cardio-metabolic health post-pregnancy is explained by pre-pregnancy subclinical cardiometabolic health. As secondary aims the study also aims to determine which aspects of pre-pregnancy cardiometabolic health impact on women's cardiovascular adaptation to pregnancy; whether haemodynamic maladaptation is an early pregnancy biomarker for the later clinical manifestations of placental dysfunction; and whether an uncomplicated pregnancy results in improved maternal cardiometabolic health post-partum. Finally, the investigators will determine whether pre-pregnancy cardiovascular risk factors affect the rate of early fetal loss (miscarriage), which will answer an important clinical question, as recurrent miscarriage is associated with increased cardiovascular risk.

ELIGIBILITY:
Pregnancy Arm Inclusion Criteria:

To be included in the trial the participant must:

* Nulliparous (no previous pregnancy beyond 20 weeks' gestation)
* Actively considering pregnancy within approximately 12 months
* Aged between 18 and 45 years
* Ability to consent and willing to participate

Pregnancy Arm Exclusion Criteria:

The presence of any of the following will preclude participant inclusion:

* Currently pregnant
* Established infertility
* Planning or actively using fertility treatments (e.g. IVF, ICSI, FET, IUI)
* Assigned male sex at birth
* Autoimmune disease (e.g. rheumatoid arthritis, lupus)
* Thrombophilia
* Type 1 diabetes
* Known advanced chronic kidney disease (stages 4-5)
* Malignant hypertension
* Clinically manifest CVD (e.g. previous myocardial infarction, stroke)
* Active cancer/being treated for cancer currently (other than skin cancer)
* Any other condition preventing full participation in the study

Non-Pregnancy Arm Inclusion criteria

To be included in the trial the participant must:

* Nulliparous (no previous pregnancy beyond 20 weeks' gestation)
* Not planning to conceive during next 18 months
* Aged between 18 and 45 years
* Ability to consent and willing to participate

Non-Pregnancy Exclusion Criteria

The presence of any of the following will preclude participant inclusion:

* Currently pregnant
* Planning or actively using fertility treatments (e.g. IVF, ICSI, FET, IUI)
* Assigned male sex at birth
* Autoimmune disease (e.g. rheumatoid arthritis, lupus)
* Thrombophilia
* Type 1 diabetes
* Known advanced chronic kidney disease (stages 4-5)
* Malignant hypertension
* Clinically manifest CVD (e.g. previous myocardial infarction, stroke)
* Active cancer/being treated for cancer currently (other than skin cancer)
* Any other condition preventing full participation in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Nulliparous women to maximise the occurrence of placental syndrome.
Sampling Method: Non-Probability Sample
Enrollment: 3500 (Estimated)
Dates: Start 2023-05-24 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2052-12 (Estimated)

PRIMARY OUTCOMES:
QRISK3 | Risk difference between women who experienced a healthy pregnancy and those who experienced a pregnancy complication at 9-12 months postpartum
  Predicted lifetime CVD risk

SECONDARY OUTCOMES:
Blood Pressure Systolic, Blood Pressure Diastolic Pulse Wave Analysis: Supine Systolic BP, Supine diastolic BP, Central Systolic BP, Central diastolic BP, Supine MAP | Assessed at 9-12 months postpartum
  BP (mmHg)
Height | Assessed at 9-12 months postpartum
  m
BMI | Assessed at 9-12 months postpartum
  kg/m2
BMR | Assessed at 9-12 months postpartum
  KJ
Waist:Hip ratio | Assessed at 9-12 months postpartum
  Waist measurement (cm), Hip measurement (cm), Waist/Hip measurement
Body fat (%), Tanita (%) | Assessed at 9-12 months postpartum
  (Tanita scales)
Weight, Fat mass, Fat free mass, Total body water | Assessed at 9-12 months postpartum
  kg
Sodium, Potassium, Urea, Total Cholesterol, Triglyceride, HDL-Cholesterol, LDL-cholesterol, Non-HDL cholesterol | Assessed at 9-12 months postpartum
  Lipids (mmol/L)
Creatinine | Assessed at 9-12 months postpartum
  Lipids (µmol/L)
HbA1c | Assessed at 9-12 months postpartum
  Lipids (mmol/mol)
White blood count (WBC), Platelet count, Neutrophil count, Lymphocyte count, Monocyte count, Eosinophil count, Basophil count | Assessed at 9-12 months postpartum
  Lipids (10*9/L)
Red blood cell (RBC) | Assessed at 9-12 months postpartum
  Lipids (10*12/L)
Haemoglobin (Hb) Haemoglobin (Hb) Haemoglobin (Hb) | Assessed at 9-12 months postpartum
  Lipids (g/L)
Haematocrit | Assessed at 9-12 months postpartum
  Lipids (L/L)
Mean cell volume (MCV) | Assessed at 9-12 months postpartum
  Lipids (fL)
Mean cell haemoglobin (MCH) | Assessed at 9-12 months postpartum
  Lipids (pg)
Red cell distribution width (RDW) | Assessed at 9-12 months postpartum
  Lipids (%)
Urine | Assessed at 9-12 months postpartum
  Protein, Blood, Glucose, Leukocytes, Nitrites
APWV: Aortic Pulse Wave Velocity, Carotid Intima-media thickness | Assessed at 9-12 months postpartum
  Suprasternal notch to distal (Femoral artery) (mm), Suprasternal notch to proximal (carotid artery) (mm), Carotid IMT (mm)
Oral glucose tolerance test (OGGT) | Assessed at 24-28 weeks pregnancy
  mmol
Diabetes Risk | Risk difference between women who experienced a healthy pregnancy and those who experienced a pregnancy complication at 9-12 months postpartum
  QDiabetes 2018

CONTACTS AND LOCATIONS:
Overall Officials: Ian Wilkinson, MD, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Cambridge University Hospitals NHS Foundation Trust, Cambridge
  - NHS Greater Glasgow and Clyde, Glasgow
  - University College London Hospitals NHS Foundation Trust, London
  - King's College Hospital NHS Foundation Trust, London
  - St George's University Hospitals NHS Foundation Trust, London
  - Imperial College Healthcare NHS Trust, London
  - Manchester University NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: Yes
Data will only be available to request after the investigator has finished with the data and will not included patient identifiable data.